CLINICAL TRIAL: NCT06211374
Title: Communication Bridge: Optimizing an Evidence-based Intervention for Individuals With Primary Progressive Aphasia
Brief Title: Communication Bridge Pilot Study
Acronym: CB3_1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Western University, Canada (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB23-1620; 7R01AG055425-07 (NIH)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Primary Progressive Aphasia
Keywords: Aphasia; Dementia; Communication; Frontotemporal Dementia; Alzheimer Disease
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia; Dementia; Communication; Frontotemporal Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Communication Bridge™ (Experimental): Participants receive Communication Bridge™, a multi-component, participation-focused, dyadic intervention in which both the person with PPA and their co-enrolled communication partner are intervention recipients. Communication Bridge™ is modelled on the Living with Aphasia: Framework for Outcome Measurement (A-FROM) and the Care Pathway Model that was developed for persons living with primary progressive aphasia. Consistent with participation-focused intervention models personally salient training stimuli are incorporated into all therapy activities in the Experimental arm.
  Interventions: Behavioral: Communication Bridge

INTERVENTIONS:
Behavioral: Communication Bridge — Evidence-based speech language therapy treatment will be compared and contrasted in the two arms of the study.

SUMMARY:
The aim of this study is to evaluate the effectiveness and feasibility of evidence-based interventions in individuals living with mild to moderate primary progressive aphasia (PPA) that address communication-focused outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness and feasibility of evidence-based interventions in individuals living with mild to moderate primary progressive aphasia (PPA) that address communication-focused outcomes. The study team aims to enhance the personal relevance and therapeutic impact of goal attainment scaling (GAS) while building self-efficacy within a self-management framework.

This study will be a continuation of one of the largest non-pharmacologic intervention studies for individuals with PPA to date. It will add critical information regarding the effectiveness of telepractice interventions for communication disorders in adults with primary progressive aphasia specifically, and in dementia more broadly. The goal of this study is to maximize functional communication and life participation for the participants.

ELIGIBILITY:
Inclusion Criteria (person with PPA):

1. Meets diagnostic criteria for PPA based on neurologist and supporting medical assessments (extracted from medical records)
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Adequate vision (aided or unaided) for reading a newspaper, or other functional materials (by self-report)
5. Able to pass technology screening and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)
6. Geriatric Depression Scale score ≤ 9
7. Mild-moderate PPA informed by a structured interview with a speech-language pathologist and a standardized testing battery.

Inclusion Criteria (Co-enrolled communication partner):

1. 18+ years of age
2. English as primary language used in daily communication activities (by self-report)
3. Adequate hearing (aided or unaided) for communicating with others in a crowded room (by self-report)
4. Able to pass technology screening* and demonstrates sufficient knowledge for use of video conference and Communication Bridge™ web application use (with or without training)

Exclusion Criteria:

* A dementia diagnosis other than Primary Progressive Aphasia
* Participation is co-enrolled in an outside speech language therapy program during the study course.
* Communication partners will be excluded if they have a pre-existing communication impairment that would affect study participation (e.g., aphasia, dementia) Medical records will be requested and reviewed to determine eligibility

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Communication Participation Person Centered Goals | Time Frame: 2 assessment time points through study completion, an average of 5 months, including change over time
  Goal Attainment Scaling, a 7-point rating scale with -3 representing 'no longer participating' and +3 representing 'exceeded goal'. Higher scores indicate better progress in goal achievement.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Roglaski, PhD, Principal Investigator — Professor of Neurology
Locations (1):
- University of Chicago - American School Building, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided